CLINICAL TRIAL: NCT07083661
Title: Mindfulness-based Intervention on Parent Empowerment in Reducing Young Children's Screen Time (MORE): a Mixed Method Study
Brief Title: Mindfulness-based Intervention and Young Children's Screen Time
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hong Kong Metropolitan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RD/2025/1.7
Record Dates: First submitted 2025-07-04; First posted 2025-07-24 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Screen Time Exposure
Keywords: screen time exposure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness-based intervention on parent empowerment in reducing children's screen time (MORE) (Experimental): The intervention consists of 6-session mindfulness-based intervention. Each session last for 2 hours. The training will be led by an experience certified mindfulness teacher.
  Interventions: Behavioral: Mindfulness-based intervention on parent empowerment in reducing children's screen time (MORE)
- Waistlist control group (No Intervention): Participants will be required to maintain their usual daily activities without begin any mindfulness and skills programme for 6-week

INTERVENTIONS:
Behavioral: Mindfulness-based intervention on parent empowerment in reducing children's screen time (MORE) — Participants will receive a 6-week MORE group training by integration of mindfulness-based component into a modified Hands-on Parent Empowerment-20 (HOPE-20) programme.
  Arms: Mindfulness-based intervention on parent empowerment in reducing children's screen time (MORE)

SUMMARY:
This research proposal aims to explore the effectiveness of the mindfulness-based intervention (MBI) on reducing young children's screen time (ST) and caring parents' psychological and social issues in Hong Kong.

DETAILED DESCRIPTION:
The research design was a two-arm waitlist, randomised controlled study with a focus group interview with 60 participants. The intervention integrates the mindfulness-based component into a modified Hands-on Parent Empowerment-20 (HOPE-20) programme, and is named as MORE (i.e. Mindfulness-based intervention On parent empowerment in REducing children's screen time). The intervention consists of 6 weeks of MBI training, each lasting for 2 hours, led by an experienced certified mindfulness teacher. The intervention programme consists of three components: (1) skill part - 4 lessons talk about parenting skills (Praising, token system, response cost, planned ignorance, quiet zone); (2) skill part - 2 lessons talk about child-parent communication (building relationship, communication strategies); and (3) mindfulness part - mindfulness-based training. The primary outcomes are young children's ST and children's disruptive behaviour. Feasibility outcomes include recruitment rate, retention rate, and acceptability of the interventions. Secondary outcomes include parent-child relationships, parents' perceptions of their abilities to manage the demands of parenting, parental stress level, and social support adequacy. The proposal also includes plans for focus group interviews with participants to gather qualitative data. Analyses will include descriptive statistics, Pearson's chi-square test, Pearson's product-moment correlations, One-way ANOVA. A p-value < 0.05 will be taken as the level of statistical significant. The 95% Confidence interval (CI) around the differences will be calculated. For qualitative data, the results will be analyzed descriptively and narratively. The proposal highlights the potential of MBI for reducing young children's ST, as well as improving children-parent relationships, enhancing the efficacy and satisfaction level of the parents, and reducing the stress level of the parents.

ELIGIBILITY:
Inclusion Criteria:

* parent-child dyads resident in Hong Kong;
* child being between 2 and 6- year; and
* child with normal intellectual ability.

Exclusion Criteria:

* children with major developmental problems, history of domestic violence, drug abuse, or mental illness in the family;
* being unable to communicate and understand Cantonese as the intervention will be conducted in Cantonese; and
* parent-child dyads previous participation in mindfulness-based training for less than 6 months.

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Screen time exposure - frequency | Baseline, week 6, week 18
  Children's screen time exposure including frequency will be record in terms of times per week
Screen time exposure - duration | Baseline, week 6, week 18
  Duration will be record in terms of minutes
Screen time exposure - nature and content | Baseline, week 6, week 18
  Screen time exposure, nature, and content require the parent to provide the types and names of the shows watched by their young children.
Screen time exposure - viewing behavior | Baseline, week 6, week 18
  The parents are required to provide the information on young children's viewing behavior, including singing, role play, discussing issues or discussing the films and shows by selecting from the questionnaire.
Change in parental stress level | Baseline, week 6, week 18
  The Parenting Stress Index - short form. It is a 36-item 5-point Likert scale with three 12-item subscales. Each item is scored from 1 to 5 (1 = "strongly disagree", 5 = "strongly agree"). The lowest score is 36, and the highest score is 180. Higher scores indicated higher parenting stress, and the cutoff point is >90.
Change in social support adquency level | Baseline, week 6, week 18
  The Multidimensional Scale of Perceived Social Support Questionnaire is a 12-item questionnaire. Each item is scored from 1 to 7 (1 = "strongly disagree", 7 = "strongly agree"), the lowest score is 12 and the highest score is 84. A higher score defines higher social support from family, friends and significant others.

SECONDARY OUTCOMES:
Change in children disruptive behavior | Baseline, week 6, week 18
  The Eyberg Child Behaviour Inventory is a 36-item questionnaire that consists of two subscales: the intensity scale and the problem scale. The intensity scale assesses the common child behavior problems frequency from 1 to 7 (1 = "never", 7 = "always"), and the problem scale assesses the extent to which the parents find the troublesome behavior in "yes" or "no". The lowest score is 36, and the highest score is 252. Higher scores indicate more child behavior problems.
Change in parent-child relationships | Baseline, week 6, week 18
  The Parenting Sense of Competence Scale is a 6-point Likert scale with 15-item. Each item is scored from 1 to 6 (1 = "strongly disagree", 6 = "strongly agree"), the lowest score is 15, and the highest score is 90. A higher score represents a better parent-child relationship

OTHER OUTCOMES:
Feasibility of the study - recruitment and retention rate | week 6, week 18
  Recruitment and retention rates will be recorded as a percentage.
Feasibility of the study - attendance rates | week 6, week 18
  Attendance rates are defined as the number of training sessions a subject has attended.
Feasibility of the study - time required to recruit to target sample size | week 6, week 18
  The time required to recruit to target sample size will be record in terms of week
Feasibility of the study - adverse events | week 6, week 18
  Adverse events will be recorded in terms of narrative style.
Acceptability of the study | week 6, week 18
  Perception and satisfaction level of the intervention programme will be assessed by questionnaire
Comments and suggestions on intervention programme | week 6, week 18
  A total of 10 parent-child dyads will be invited to an hour focus group interview after the completion of the MORE programme to gather the experiences of participants.
  A semi-structured interview question will be used for focus group discussions and individual interviews, and an audio recorder will be used to record the dialogue of the focus group interview. The audiotaped interviews will be transcribed verbatim by a trained RA.

CONTACTS AND LOCATIONS:
Overall Officials: Yuen Ling Leung, Doctor of Nursing, Principal Investigator — Hong Kong Metropolitan University

IPD SHARING:
Plan to Share IPD: No